CLINICAL TRIAL: NCT07240155
Title: COMPARATIVE EFFICACY OF OZONE INJECTIONS AND HOME-BASED EXERCISE ON LATERAL EPICONDYLOPATHY
Brief Title: Ozone Therapy in Lateral Epicondylopathy
Acronym: O2-O3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: Izmir Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Demir Benli, Medical Doctor, Dokuz Eylul University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Atatürk Education and Research
Record Dates: First submitted 2024-07-19; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Tennis Elbow
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ozone (Experimental): The ozone therapy sessions were applied while the patient was in the supine position. The location and depth of the injection points were identified through palpation. Povidone iodine has been used for sterilization. The injection site was cleaned in accordance with the aseptic antisepsis guidelines. The injection was applied at trigger points. First, the lateral epicondyle was determined and marked and then trigger points were determined and marked. After the skin was sterilized, injections were made using a 25-gauge 1.5-inch needle without applying local anesthesia to lateral epicondyle with 90° elbow flexion. In each session, 5-7 ml, 15μg/mL O2-O3 in trigger points for each region according to the Unification of Criteria in the Practice of Ozone Therapy (as described in the Madrid Declaration). Ozon injections were performed six times at 3-4 day intervals
  Interventions: Device: Ozone treatment

INTERVENTIONS:
Device: Ozone treatment — tThe home-based exercise consisted of streching, strenghtening for wrist and elbow. Participants implemented the home exercise program once a day, every day of the week.
  Other Names: home-based exercise therapy

SUMMARY:
Lateral epicondylopathy (LE) is a common cause of elbow pain. In the literature, there are few studies evaluating the efficacy of ozone injection in LE. To our knowledge, there is no study comparing it with exercise therapy. This study aims to investigate the efficacy of home-based exercise and ozone therapy on pain, functionality and quality of life in LE.

DETAILED DESCRIPTION:
Introduction: Lateral epicondylopathy (LE) is a common cause of elbow pain. In the literature, there are few studies evaluating the efficacy of ozone injection in LE. To our knowledge, there is no study comparing it with exercise therapy. This study aims to investigate the efficacy of home-based exercise and ozone therapy on pain, functionality and quality of life in LE. A rehabilitation hospital associated with a community-based tertiary medical center. In this study, 65 patients with clinically diagnosed LE received either home-based exercise (Group 1), ozone injections (Group 2). Data from 59 patients were analyzed.

ELIGIBILITY:
Inclusion criteria were that the patients' age was ranged from 18 to 65, they were diagnosed with lateral epicondylitis, and they received ozone or exercise therapy, and had sufficient data.

Exclusion criteria consisted of any injections for LE within last six months, arthritis, effusion around the elbow, infection or trauma involving lateral epicondylar region, any previous fractures of the forearm or upper arm, physiotherapy within last six months, deformities or neurological deficits of the upper extremity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | VAS values were measured before treatment, one month and three months after treatment.
  All the patients were examined for pain of elbow using a Visual Analog Scale (VAS) that rated the severity of pain on a scale of 0 to 10, where 0 indicated no pain and 10 signified severe pain.
Patient-rated Tennis Elbow Evaluation (PRTEE) | PRTEE values were measured before treatment, one month and three months after treatment.
  PRTEE is a valid outcome measure for rating pain (PRTEE-pain) and disability (PRTEE-function) for forearm, that specifically developed for patient with LE. The scale has two parts, for pain (5 items) and function (10 items). Each item has a score from 0 to 10; a score of 10 refers to severe pain or inability to perform the activity.
Quick Disabilities of the Arm, Shoulder and Hand (Quick-DASH) | Quick-DASH values were measured before treatment, one month and three months after treatment.
  Quick-DASH questionnaire evaluates upper extremity disability levels. Quick-DASH contains 11 items (scored 1-5) that evaluate the daily living activities and severity of symptoms. A higher score indicates greater disability.

SECONDARY OUTCOMES:
European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3L) | EQ-5D-3L values were measured before treatment, one month and three months after treatment.
  The EQ-5D-3L descriptive system consists of the following five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has three levels: no problem (1 point), some problem (2 point), and extreme problem (3 point). The EQ-VAS records the patient's self-rated health on a vertical VAS where ranged from 0 (worst imaginable health state) - 100 (the best imaginable health state).

CONTACTS AND LOCATIONS:
Locations (1):
- Merve Demir Benli, Izmir, Balçova, Turkey (Türkiye)